CLINICAL TRIAL: NCT05880511
Title: Augmented Reality Sensorimotor Training to Treat Chronic Neck Pain Assessed Through Corticomuscular Coherence
Brief Title: Augmented Reality Sensorimotor Training to Treat Chronic Neck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16310
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Sham) (Sham Comparator): Participants in group A will take part in 2-4 weeks of treatment with 3-5 sessions per week. Each session will involve both sham repetitive transcranial magnetic stimulation (rTMS) and augmented reality sensorimotor training. Sham repetitive transcranial magnetic stimulation (rTMS) will be delivered at 10 Hz, 2000 pulses targeting the hand representation of the left primary motor cortex. Participants will hear and experience the clicking but will not be provided with any stimulation. Sham rTMS will take approximately 11.5 minutes. Immediately following sham rTMS, participants will perform augmented reality sensorimotor training. Participants will perform 20 minutes of sensorimotor training.
  Interventions: Device: Augmented Reality Sensorimotor Training; Device: Sham Repetitive transcranial magnetic stimulation
- Group B (Active) (Experimental): Participants in group B will take part in 2-4 weeks of treatment with 3-5 sessions per week. Each session will involve both real repetitive transcranial magnetic stimulation (rTMS) and augmented reality. Repetitive transcranial magnetic stimulation (rTMS) will be delivered at 10 Hz, 2000 pulses targeting the hand representation of the left primary motor cortex. rTMS will take approximately 11.5 minutes. Immediately following rTMS, participants will perform augmented reality sensorimotor training. Participants will perform 20 minutes of sensorimotor training.
  Interventions: Device: Repetitive transcranial magnetic stimulation; Device: Augmented Reality Sensorimotor Training

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. 2000 pulses will be delivered at 10 Hz stimulation. Stimulation will be delivered at 80% of the resting motor threshold obtained from the right APB muscle. The delivery of rTMS requires ~ 11.5 minutes in total.
  Other Names: rTMS, Repetitive TMS
  Arms: Group B (Active)
Device: Augmented Reality Sensorimotor Training — Sensorimotor training is a non-invasive, non-painful procedure using augmented reality to present virtual objects which cue motor action. Augmented reality allows us to project virtual objects overlaid on the user's actual environment. The sensorimotor training task involves making movements with the head and neck such that a target crosshair presented in the centre of the glasses is moved to a virtual target that is presented in the user's environment. Participants will perform 20 minutes of sensorimotor training. The goal of augmented reality sensorimotor training is to promote goal directed actions using the head and neck.
Device: Sham Repetitive transcranial magnetic stimulation — Sham repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, non-painful procedure. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. During the sham, participants will hear and experience the clicking from the device but will not be provided with any stimulation. The delivery of sham rTMS requires ~ 11.5 minutes in total.
  Arms: Group A (Sham)

SUMMARY:
The goal of this research is to investigate whether 2-4 weeks of augmented reality sensorimotor training induces positive changes so as to effect pain relief in patients with chronic neck pain. In addition, this study aims to determine if repetitive transcranial magnetic stimulation (rTMS) delivered prior to augmented reality sensorimotor training enhances the benefits from the sensorimotor training. This study will also use a battery of questionnaires, functional assessments and electroencephalography markers to identify changes following the sensorimotor training that may be associated with benefits in pain symptoms. Before we embark on a larger study, we plan to investigate the feasibility of our study procedures in a feasibility study involving 40 patients.

DETAILED DESCRIPTION:
Chronic neck pain (CNP) is cervical pain that arises in the absence of a traumatic injury or other known pathological abnormality (Borghouts et al., 1998; Cerezo-Téllez et al., 2016). CNP is associated with deficits in motor control (Jull & Falla, 2016), increased fatiguability (Falla et al., 2003), and hyperalgesia, such as increased pain sensitivity to pressure and heat (Castaldo et al., 2019; Piña-Pozo et al., 2019). Patients with CNP also experience myofascial pain syndrome (Cerezo-Téllez et al., 2016; Fernández-de-las-Peñas et al., 2007). Myofascial pain syndrome is referred pain from myofascial trigger points that can cause autonomic, sensory, and motor effects in areas distant from the trigger point (Cerezo-Téllez et al., 2016). CNP is a debilitating condition that leads to decreased quality of life and affects approximately 22% of Canadians (Côté et al., 1998). Previous work has cited that the incidence of CNP increases with age (Andersson et al., 1993; Brattberg et al., 1989; McLean et al., 2010). Individuals aged 45-55 are twice as likely to develop CNP compared to younger individuals (Korhonen et al., 2003). Age is also associated with poorer pain outcomes at 3 and 12 months following the arise of symptoms (Bot et al., 2005). Despite this, no gold standard treatment for older individuals with CNP currently exists.

Recently, virtual reality has been used to treat pain and motor symptoms of CNP. Specifically, this approach works by promoting goal directed movements of the neck towards targets presented within a virtual environment. Neck training using virtual reality (VR) has been shown to be as effective as manual exercise for improving pain and mobility in individuals with chronic neck pain (Tejera et al., 2020; Grassini 2022). In addition, VR may be more engaging compared to traditional exercise and shows an additional improvement in proprioception, pain, and decreased functional limitations (Cetin et al., 2022) beyond traditional exercise (Nusser et al., 2021). These environments also distract participants with CNP from pain during movements aiming to positively influence kinesiophobia (Luque-Suarez et al., 2019). Additionally, these effects have been suggested to occur as a result of increased eye-head coordination required to successfully navigate and interact with object within the VR environment (Revel et al., 1994: Humphreys & Irgens 2002) which promotes neural connectivity between the vestibular system, neck, and eyes (Sarig et al., 2015). These environments can also be adaptable to participant performance and require complex and dynamic movements to complete certain tasks. These movements may improve an individual's perception of cervical position and fine motor control which has been shown to lead to a reduction in neck pain symptoms (Jull et al., 2007; Röijezon et al., 2008). We have developed a novel augmented reality (AR) sensorimotor training task that promotes targeted goal directed actions with the head and neck. AR is defined as technology that overlays digital object or information into the real world (Berryman 2012). AR provides a unique opportunity for participants to engage in training that may benefit sensorimotor control of neck movements. Specifically, it allows for users to interact with virtual object overlaid on their actual environment.

The beneficial effects of AR training may indeed be enhanced using repetitive transcranial magnetic stimulation (rTMS) prior to AR training. Specifically, rTMS delivered to the primary motor cortex may create an environment within the sensory motor cortex that promotes neuroplasticity. This is accomplished through high frequency rTMS which increase cortical excitability (León et al., 2018). This in turn promotes intraneuronal connectivity and reorganization achieved through sensorimotor integration provided by the AR sensorimotor training task. Additionally, rTMS facilities neuroplasticity and the retraining of cortical circuits. This can be used to restore cortical activity that is altered in patients with CNP (León et al., 2018).

Changes to the primary motor cortex (M1) have been implicated in the pain network underpinning CNP. These include changes in the cortical territory (Elgueta-Cancino et al., 2019) and activation patterns of the area representing the affected muscles during painful and non-painful head movements (Beinert et al., 2017). Additionally, increased resting state functional connectivity between M1 and superior parietal cortex has been associated with greater local hyperalgesia (Coppieters et al., 2021). Taken together, these results suggest altered sensorimotor processing during motor control of the neck leads to pain. This is supported by findings in subclinical neck pain that have demonstrated deficits in neuromuscular control of the neck (Zabihhosseinian et al., 2015), sensorimotor processing (Baarbé et al., 2016), sensorimotor integration, and greater inhibition of the motor cortex (Baarbé et al., 2018) in patients with subclinical neck pain compared to healthy controls. As a result, changes in sensorimotor control between the cortex and affected muscles may accompany changes in pain symptoms following a sensorimotor training intervention. Sensorimotor control in CNP may be reflected in corticomuscular coherence (CMC). CMC is derived from the correlation between electroencephalography recorded over the primary motor cortex and electromyography recorded from an active muscle. CMC is suggested to reflect the flow of information from the motor cortex to the muscle, as well as feedback from the muscle back to the somatosensory cortex (Gross et al., 2000; Lim et al., 2014; McClelland et al., 2012; Riddle & Baker, 2005; Salenius et al., 1997; Witham et al., 2011). In healthy participants, von Carlowitz-Ghori et al. (von Carlowitz-Ghori et al., 2015) demonstrated that CMC can be volitionally modified. During a steady state hold with the thumb, participants improved their CMC value through different strategies such as mental imagery and attention (von Carlowitz-Ghori et al., 2015). Taken together, these results suggest that CMC can reflect deficits in cortical control of movement and may be used as a marker of improved sensorimotor control between the brain and active muscle following a training task implemented using AR.

The objective of our study is to investigate the use of rTMS paired with a novel AR sensorimotor training task in CNP patients, to induce positive neuroplastic changes so as to effect temporary and long-term pain relief. In addition, this study aims to determine if AR leads to improvements in sensorimotor control of the neck measured through CMC. AR sensorimotor training may induce cortical reorganization and improve motor function leading to analgesic effects in patients with CNP. In addition, this is the first study in CNP to use CMC to assess deficits observed in the voluntary sensorimotor control of muscles of the neck.

Effective long-term pain relief for older patients with CNP is currently an unmet medical need. As such, this work aims to implement an innovative technique to provide meaningful and long-lasting pain relief. This intervention aims to break the cycle of pain and improve activities of daily living and quality of life in CNP. This is the first study to the best of our knowledge combing rTMS with AR to treat patient with CNP.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of chronic neck pain

Exclusion Criteria:

* A known history of moderate to severe chronic pain in other parts of the body
* Contraindications to transcranial magnetic stimulation,
* Known psychological diagnosis affecting comprehension
* Inability to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability to recruit 20 patients in each group over a 6-month period | Immediately following the intervention.
  Ability to recruit 20 patients in each group over a 6-month period
Compliance of treatment sessions for the two groups | Immediately following the intervention.
  Compliance of sessions is defined as a minimum of attending 3 sessions per week for 2 weeks.

SECONDARY OUTCOMES:
PROMIS-29 v2.0 Profile | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  Using numerical rating (0 to 5) to assess seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Also uses a numerical rating to asses pain intensity (0-10).
Visual analog scale | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  A 10 cm straight line that is marked in order to indicate the severity of pain. The left edge fo the line is considered no pain at all and the right edge is considered the worst pain possible.
Pressure pain threshold (PPT) | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  Used to measure deep muscular tissue sensitivity. Pressure is applied to a given areas and is steadily increased until it turns into a painful pressure sensation
Patient Perceived Global Index of Change (PGIC) | Immediately following intervention, 2 weeks after intervention
  1-7 Likert Scale: Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse
The neck disability index | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  A 10-item questionnaire used to measure self-rated disability due to neck pain
Tampa Scale of Kinesiophobia | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  A 17-item questionnaire used to quantify fear of movement. Each question is scored from 1 (strongly disagree) to 4 (strongly agree). The total score ranges from 11-44 points with higher scores indicating greater fear of pain, movement, and injury.
Non-Likert type enjoyment scale | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  A 4 point scale used to measure how much participants enjoyed the study intervention. Higher scores are related to more enjoyment and lower scores related to less enjoyment.
Active cervical range of movement (CROM) | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  Assessed using the CROM device. This device consists of two goniometers that are used to measure range of motion during different planes of movement. This device has been verified to be reliable for measuring cervical ROM.
Augmented Reality Time to Target | Through study completion
  Performance metric data is recorded during the augmented reality sensorimotor training through accelerometers built into the augmented reality glasses. This metric specifically measures the amount of time it takes for participants to complete the targeted action during sensorimotor training. Higher time to target scores represent worse outcome and lower scores represent better performance.
Motor evoked potential recruitment curve | 2 week before intervention, immediately before intervention, immediately following intervention, 2 weeks after intervention
  This TMS measure will involve stimulating the motor hotspot for the abductor pollicis brevis muscle with single pulses ranging from 90% of resting motor threshold (RMT) to 150% RMT. This measure is performed to determine if any excitability changes have occurred as a result of the rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Nelson, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton King Campus, Hamilton, Ontario
  - McMaster Unviersity, Hamilton, Ontario